CLINICAL TRIAL: NCT02623439
Title: A Phase 2 Study of Nonmyeloablative Conditioning With Transplantation of Partially Human Leukocyte Antigen (HLA)-Mismatched Bone Marrow and Post-transplant Cyclophosphamide for Patients With Hematologic Malignancies
Brief Title: A Study of Haploidentical Bone Marrow Transplant for Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Caitlin Costello, MD, Assistant Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120931
Record Dates: First submitted 2013-08-29; First posted 2015-12-07 (Estimated); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
Keywords: hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cyclophosphamide post BMT (Experimental): Cyclophosphamide 50 mg/kg IV Days 3 and 4 post transplant
  Interventions: Drug: Cyclophosphamide 50 mg/kg IV Days 3 and 4 post transplant

INTERVENTIONS:
Drug: Cyclophosphamide 50 mg/kg IV Days 3 and 4 post transplant — Cyclophosphamide 50 mg/kg IV Days 3 and 4 post transplant

SUMMARY:
The primary objective is to determine overall survival 180 days after transplantation involving HLA-haploidentical stem cell/bone marrow graft, and post-transplant Cy.

DETAILED DESCRIPTION:
Study Design: This is a single center Phase 2 study of myeloablative (MA) and nonmyeloablative (NMA) conditioning, transplantation of partially HLA-mismatched bone marrow or peripheral blood stem cells and post-transplantation cyclophosphamide (Cy) in patients with hematologic malignancies including:

1. Acute lymphoblastic leukemia/lymphoma, acute myelogenous leukemia, and Burkitt's lymphoma in remission.
2. Relapsed lymphoma, including marginal zone B cell lymphoma, follicular lymphoma, and chemotherapy-sensitive large-cell or Hodgkin lymphoma.
3. Myelodysplastic Syndrome (MDS)
4. Blastic plasmacytoid dendritic cell neoplasm

Primary Objective:

The primary objective is to determine overall survival 180 days after transplantation involving Myeloablative and Non myeloablative conditioning, HLA-haploidentical marrow or peripheral blood stem cell grafts, and post-transplant Cyclophosphamide as GVHD prophylaxis.

Secondary Objectives:

Secondary objectives include estimating overall and progression-free survival at 100 days, 180 days, and one year after transplantation, treatment-related mortality, incidence of neutrophil and platelet recovery or engraftment, incidence of graft failure, cumulative incidence of acute and chronic Graft versus Host Disease (GVHD), incidence of infections, and cumulative incidence of relapse/progression. The investigators will also examine the amount of time to transplant (day of unrelated search initiation to day 0).

ELIGIBILITY:
Inclusion Criteria:

1. Age: Subjects 18-70 years old.
2. Donor must be 18 years of age.
3. HLA typing will be performed at high resolution. A minimum match of 5 out of 10 is required.
4. Patients must have received multi-agent chemotherapy within 3 months of consent date (measured from the start date of chemotherapy).
5. Acute Leukemias.

   * Acute Lymphoblastic Leukemia in high risk 1st complete response (CR1)
   * Acute Myelogenous Leukemia in high risk 1st complete response (CR1)
   * Acute Leukemias in 2nd or subsequent Complete Response (CR)
   * Biphenotypic/Undifferentiated Leukemias in 1st or subsequent Complete Response (CR).
6. Burkitt's lymphoma: second or subsequent Complete Response (CR).
7. Lymphoma
8. Patients with adequate physical function
9. Performance status: Karnofsky score 70-100%.

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09-21 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Caitlin, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | cyclophosphamide post BMT
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide Post BMT
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: 180 days after transplantation
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | cyclophosphamide post BMT
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | cyclophosphamide post BMT
All-Cause Mortality (participants affected / at risk) | 5/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cyclophosphamide post BMT (N=8)
Renal Failure (Renal and urinary disorders) | 1 (1)
CMV (Immune system disorders) | 1 (2)
Adenovirus (Immune system disorders) | 1 (1)
Acute GVHD (Immune system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cyclophosphamide post BMT (N=8)
Human herpesvirus 6 (HHV-6) (Immune system disorders) | 1 (2)
Enterococcus Faecalis UTI (Infections and infestations) | 1 (1)
BC (+) Rothia mucilaginosa septicemia (Infections and infestations) | 1 (1)
CMV (Immune system disorders) | 1 (1)
acute GVHD (Immune system disorders) | 2 (3)
aspergillosis (Immune system disorders) | 1 (2)
stenotrophomomas pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cytokine storm (Blood and lymphatic system disorders) | 2 (2)
vancomycin-resistant enterococcus (VRE) (Infections and infestations) | 1 (1)
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
extended spectrum beta-lactamase (ESBL) E.Coli (Infections and infestations) | 1 (1)
Systemic inflammatory response syndrome (SIRS) (Infections and infestations) | 1 (1)
Clostridioides difficile or C-diff (Infections and infestations) | 2 (2)
CMV viremia (Immune system disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02623439/Prot_SAP_000.pdf